CLINICAL TRIAL: NCT05432921
Title: Evaluation of Outpatient Cardiac Rehabilitation in Austrian Outpatient Facilities.
Brief Title: Cardiac Rehabilitation in Austrian Outpatient Facilities.
Acronym: EvOCaReAustria
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Prof. Josef Niebauer M.D., Ph.D., MBA (Other)
Responsible Party: Sponsor-Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Head of Institute, Paracelsus Medical University
Organization: Paracelsus Medical University (Other)
Other Study IDs: UISM-15
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases
Keywords: cardiac rehabilitation; exercise training; lifestyle modification; coronary-artery-disease; myocardial infarction
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lifestyle modification — 50min of endurance combined with 50min of strength training; 1-2 sessions/week for 6 month, follow up after 3-6month

SUMMARY:
Cardiac rehabilitation (CR) is a key component of the treatment of cardiac diseases. The Austrian outpatient CR model is unique, as it provides patients with an extended professionally supervised, multidisciplinary program of 4-6 weeks of phase II (OUT-II) and 12 months of phase III (OUT-III) CR CR including a "refresher". The aim of this retrospective analysis is to pool data from preferably all Austrian outpatient rehabilitation facilities and to analyze the efficacy of the Austrian cardiac rehabilitation model with a special focus on phase III. Data of patients who completed OUT-III between 1.1.2019 and 01.07.2022 will be analyzed. All patients undergo assessment of anthropometry, resting blood pressure, lipid profile, fasting blood glucose, exercise capacity, quality of life, anxiety and depression at the beginning (T1), in the middle (T2) and end of CR (T3).

DETAILED DESCRIPTION:
Cardiac rehabilitation (CR) is a multidisciplinary therapeutic intervention aimed at regaining and maintaining long-term professional and social integration. Specialist societies classify cardiac rehabilitation with the highest recommendation level (Class I). The focal points of therapy in cardiac rehabilitation include health education, optimization of risk factors through psycho-social counseling and structured physical training.

The four-tier Austrian model of cardiac rehabilitation consists of phase I, which takes place in the acute care hospital directly after a cardiac event or intervention/surgery. Phase II ideally follows immediately and lasts 3-4 weeks as an inpatient or alternatively 6 weeks as an outpatient CR. In the subsequent phase III patients ideally transfer knowledge and skills gained during rehabilitation into their daily lives. Supervised outpatient training is carried out once or twice a week for 6 months and takes part in psycho-social and physical health training courses. This is followed by a 3-6 months lasting "home phase" in which patients to follow the agreed-on lifestyle changes on their own, while documenting successes and problems. After this home phase, the Austrian model provides a "refresher" consisting of two guided outpatient training sessions as well as psychological consultation and a medical examination including a stress test. The refresher must be completed within a maximum of four weeks and is a unique feature of the Austrian model, aiming to achieve sustainable lifestyle modification. The patient-financed and life-long phase IV begins no later than 18 months after the start of phase II. Its aim is to achieve an improvement in the prognosis through lifelong, autonomous and self-responsible behavior and long-term prevention.

The aim of this retrospective analysis is to pool data from preferably all Austrian outpatient rehabilitation facilities and to analyze the efficacy of the Austrian cardiac rehabilitation model with a special focus on phase III.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who meets inclusion criteria for outpatient cardiac rehabilitation in Austria

Exclusion Criteria:

* Patients are excluded, if they don't meet the inclusion criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that completed in- our outpatient phase II and phase III out-patient cardiac rehabilitation. Diagnoses that qualify for cardiac rehabilitation paid by health insurances comprise acute coronary syndrome; percutaneous coronary intervention; stable coronary heart disease; aortocoronary bypass surgery; other surgeries of the heart and the big vessels; heart and lung transplantation; chronic heart failure; pulmonary hypertension; peripheral artery occlusive disease; prevention in motivated high risk patients; electro-physiological intervention; implantation of a cardiac pacemaker or a defibrillator; haemodynamically stable arrhythmia; sustained ventricular tachycardia or cardiac arrest.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in physical work capacity (PWC) in phase III rehabilitation | 12months
  PWC is measured during a graded exercise test on a cycle ergometer at begin and end of outpatient cardiac rehabilitation
Change from baseline in physical work capacity (PWC) within the first 6month of Phase III | 3-6months
  PWC is measured during a graded exercise test on a cycle ergometer at begin and midtime of outpatient cardiac rehabilitation

SECONDARY OUTCOMES:
Change from baseline in LDL-Cholesterol in Phase III rehabilitation | 12months
  Venous blood samples are drawn to assess Cholesterol at the start and end of Phase III rehabilitation
Change from baseline in Triglycerides in Phase III rehabilitation | 12months
  Venous blood samples are drawn to assess Triglycerides at the begin and end of Phase III
Change from baseline in Glucose in Phase III rehabilitation | 12months
  Venous blood samples are drawn to assess Triglycerides at the begin and end of Phase III

CONTACTS AND LOCATIONS:
Overall Officials: Josef Niebauer, MD, PhD, MBA, Study Director — Paracelsus Medical University
Locations (1):
- Institute of Sports Medicine, Prevention and Rehabilitation, Paracelsus Medical University, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams V, Reich B, Uhlemann M, Niebauer J. Molecular effects of exercise training in patients with cardiovascular disease: focus on skeletal muscle, endothelium, and myocardium. Am J Physiol Heart Circ Physiol. 2017 Jul 1;313(1):H72-H88. doi: 10.1152/ajpheart.00470.2016. Epub 2017 May 5. PMID 28476924
- [Result] Reich B, Benzer W, Harpf H, Hofmann P, Mayr K, Ocenasek H, Podolsky A, Pokan R, Porodko M, Puelacher C, Sareban M, Traninger H, Ziegelmeyer W, Niebauer J. Efficacy of extended, comprehensive outpatient cardiac rehabilitation on cardiovascular risk factors: A nationwide registry. Eur J Prev Cardiol. 2020 Jul;27(10):1026-1033. doi: 10.1177/2047487319898958. Epub 2020 Jan 14. PMID 31937125
- [Result] Niebauer J, Mayr K, Harpf H, Hofmann P, Muller E, Wonisch M, Pokan R, Benzer W. Long-term effects of outpatient cardiac rehabilitation in Austria: a nationwide registry. Wien Klin Wochenschr. 2014 Mar;126(5-6):148-55. doi: 10.1007/s00508-014-0527-3. Epub 2014 Mar 11. PMID 24615677
- See also: Paracelsus Medical University — http://www.pmu.ac.at
- See also: Institute of Sports Medicine, Prevention and Rehabilitation — http://www.salk.at/sportmedizin.html